CLINICAL TRIAL: NCT00859859
Title: Vagus Nerve Stimulation in Rheumatoid Arthritis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The protocol was terminated early (prior to complete enrollment) after interim analysis proved data to be statistically insignificant
Sponsor: Northwell Health (Other)
Responsible Party: Kevin J. Tracey. MD, The Feinstein Institute for Medical Research
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCRC 0137
Record Dates: First submitted 2009-03-10; First posted 2009-03-11 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Vagus Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Vagus Nerve Stimulation — 1. Vagus nerve stimulation for 5 minutes with an oscillatory device (Brookstone) used in previous experimental animal studies for stimulating the vagus nerve on the neck by carotid massage. The oscillatory part of this pen-like device is approximately 0,5 cm2.
  2. Basic lab tests (metabolic panel and CBC with differential) and monocyte cytokine synthesis and other inflammatory markers will be analyzed.

SUMMARY:
The purpose of this study is to examine the short-term effects of vagus nerve stimulation (VNS) by auricular stimulation (stimulation of the auricular branch of the vagus nerve which innervates the ear) in rheumatoid arthritis (RA). RA is characterized by a chronic systemic inflammation affecting the joints but also carries an increased risk for extra-articular manifestations as well as other organ manifestations such as cardiovascular disease (CVD), which significantly contributes to morbidity and mortality in this disorder.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a diagnosis of RA based on the ACR guidelines. Disease activity measured as activity score (DAS-28 CRP) will be used
2. None of the exclusion criteria (see below).

Exclusion Criteria:

1. Minors (<18 years of age) and mentally incompetent individuals
2. One or more of the following conditions: immunosuppressive condition (which includes malignancy, chronic alcoholism, diabetes), severe chronic dementia, psychiatric illness with active psychosis, current intravenous or other serious illicit drug use
3. Pregnancy
4. Terminal status referred for palliative care only
5. Homeless status
6. IDDM and NIDDM patients will not be enrolled in this study
7. Previous history of ischemic cardiovascular disease including myocardial infarction, unstable angina, and bradytachyarrythmias
8. Moderate or severe anemia. Hemoglobin levels will be determined at screening. A cut-off level of < 10 mg/dL in women and < 11 mg/dL in men is selected.
9. Smoking
10. Subjects taking concomitant medications potentially affecting autonomic function such as anti-cholinergic medications and beta-blockers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2006-10; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Assessment of short-term and medium-term effects of vagus nerve intervention with endpoints such as autonomic function, cytokine synthesis, inflammatory markers as well as disease activity score and global health measurement in subjects | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Kevin J Tracey, MD, Principal Investigator — Northwell Health
Locations (1):
- The Feinstein Institute for Medical Research, Manhasset, New York, United States

REFERENCES:
- [Derived] Addorisio ME, Imperato GH, de Vos AF, Forti S, Goldstein RS, Pavlov VA, van der Poll T, Yang H, Diamond B, Tracey KJ, Chavan SS. Investigational treatment of rheumatoid arthritis with a vibrotactile device applied to the external ear. Bioelectron Med. 2019 Apr 17;5:4. doi: 10.1186/s42234-019-0020-4. eCollection 2019. PMID 32232095